CLINICAL TRIAL: NCT06774794
Title: Precision Medicine in the Management of the Heart Transplant Patient: Advanced Molecular and Imaging Approaches
Brief Title: Precision Medicine in the Management of Heart Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Precision-HT; RC-2022-2773280 (Other Grant/Funding Number: Bando RC 2022-2024, Ministero della Salute)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood samples, from which cfDNA will be extracted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to demonstrate that a multiparametric approach, based on the integration of biomolecular, histological, imaging, and clinical information, along with the use of machine learning methods, can identify among heart transplant patients those at higher risk of rejection, infectious events, and chronic graft dysfunction.

Patients have been and will be treated according to clinical practice, in accordance with the physician's judgment and the information provided in the Technical Data Sheet of each individual product used in concomitant therapies, if administered according to clinical practice. The diagnostic-therapeutic pathway of the patients will not be in any way influenced by the results of tissue tests performed for the purposes of the study

DETAILED DESCRIPTION:
The main focus of the study, and the primary outcome measure, is the diagnosis of rejection based on the histopathological examination of myocardial biopsies. At the time of each biopsy procedure, or within the 5 days immediately preceding, enrolled patients will undergo specific non-invasive investigations, along with baseline clinical and laboratory evaluations.

Additional analyses will be performed on myocardial tissue samples obtained during biopsies conducted for clinical practice, including the analysis of the intramyocardial gene expression profile (nanostring and microarray), to identify molecular profiles specific to cellular or antibody-mediated rejection.

The results of these investigations will be correlated with the findings from histopathological and molecular analyses of the biopsies using artificial intelligence methods, in order to develop a non-invasive investigation algorithm that can predict the risk of rejection.

Similarly, these diagnostic investigations will be longitudinally related to the incidence of infection events, as defined above, and to the development of myocardial fibrosis diagnosed by cardiac magnetic resonance imaging.

In a subsequent phase, biopsies will be reclassified through the examination of histopathological morphology using machine learning techniques. The result of the re-evaluation of the histological samples will be correlated with the diagnosis based on the intramyocardial gene expression and the predictiveness of the previously developed algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Have received an orthotopic heart transplant
* Clinical indication for performing a myocardial biopsy (either as part of standard monitoring or for suspected rejection)
* Obtaining informed consent

Exclusion Criteria:

* Severe complications in the post-operative phase that may limit the patient's short-term survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing orthotopic heart transplantation, attending the SSD Heart Failure and Transplants unit of the IRCCS Azienda Ospedaliero-Universitaria di Bologna, will be enrolled from 01/02/2023 to 31/12/2027. Each patient will be followed according to standard clinical care practices; the minimum follow-up for each patient will be 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Histological diagnosis of rejection leading to a change in immunosuppressive therapy according to clinical practice. | 5 years
  Histological diagnosis

SECONDARY OUTCOMES:
Symptomatic infection requiring treatment with antimicrobial drugs | 5 years
  Infection from SARS-CoV-2 is excluded from this endpoint and will be analyzed separately
Development of myocardial fibrosis diagnosed on cardiac MRI | 5 years
  myocardial fibrosis diagnosis
Hospitalization for any cause. | 5 years
  Hospitalization
Mortality from any cause. | 5 years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Luciano G Potena, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Luciano, Bologna, Italy